CLINICAL TRIAL: NCT01157949
Title: A Randomized Study to Assess the Effect and Safety Profile of Thymoglobulin® for the Prevention of Cardiac Allograft Vasculopathy in Primary Cardiac Transplant Recipients: A 12-month, Single Center, Randomized, Open-label Study of Efficacy Comparing Immediate Treatment With and Without Thymoglobulin® 1.5 mg/kg/d for 5 Consecutive Days in Heart Transplant Recipients.
Brief Title: A Study to Compare the Effectiveness of a Drug That Suppresses the Immune System Called Thymoglobulin® in Preventing the Development of a Disease That Affects the Majority of Heart Transplant Recipients Called Cardiac Allograft Vasculopathy (CAV)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: PI not planning to pursue this study and it was never IRB approved.
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Jon Kobashigawa, Associate Director, Cedars-Sinai Heart Institute, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-1007-1
Record Dates: First submitted 2010-07-07; First posted 2010-07-08 (Estimated); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Cardiac Allograft Vasculopathy
MeSH Terms: interventions — thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- Study withdrawn (Active Comparator): Study withdrawn
  Interventions: Drug: Thymoglobulin
- Withdrawn (Placebo Comparator): Study withdrawn
  Interventions: Drug: Thymoglobulin

INTERVENTIONS:
Drug: Thymoglobulin — Study patients will receive 1.5 mg/kg/day intravenously for 5 days.

SUMMARY:
The purpose of this study is to test the hypothesis that administering Thymoglobulin® induction therapy early after transplant prevents the development of cardiac allograft vasculopathy (CAV). CAV accounts for a significant number of deaths in cardiac recipients after the first year of transplant. At 5 years post-transplant 30% of the deaths are due to CAV. With the exception of re-transplantation the available treatments for CAV are only effective at inhibiting its progression.

CAV involves only the allograft and spares the native arteries, suggesting an immunologic basis for the disease. However, both immunological and non-immunological factors contribute to the development of CAV. The established immunological risk factors are recurrent rejection and humoral/antibody-mediated rejection (AMR). Non-immunological risk factors identified include preservation injury, the cause of donor death, donor graft ischemic time, and cytomegalovirus infection1. It is hypothesized that these factors increase the risk of developing CAV by causing early endothelial damage to the graft, which then could promote increased lymphocyte-endothelial interactions and the production of anti-endothelial antibodies2. The investigators hypothesized that Thymoglobulin induction therapy would prevent the development of CAV because its polyclonal nature allows Thymoglobulin to target all the potential mechanisms that contribute to the development of CAV-T-cell activation, B-cell activation, antibody formation, induction of tolerance, and modulation of lymphocyte-endothelium interactions3. Because the mechanism by which Thymoglobulin affects the immune system are still poorly understood, the investigators will also study how Thymoglobulin changes the immune system over time in the heart transplant recipient as a secondary objective.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be undergoing their first allograft transplant
* Men and non-pregnant women must be 18 to 70 years old
* Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to transplantation. The sensitivity must be equal to at least 50 mIU/mL. (Urine test is allowed in addition to serum test in patients where serum results are delayed).
* Women of childbearing potential must use two reliable forms of contraception simultaneously. Effective contraception must be used before beginning study drug therapy, and for 4 months following discontinuation of study drug therapy.
* Subjects must be willing and be capable of understanding the purpose and risks of the study and must sign a statement of informed consent.

Exclusion Criteria:

* Previous organ transplants
* Patients receiving multiple organs
* Patients > 250 lbs or 114 kgs
* Patients requiring VAD upon completion of transplantation surgery. [Patients who require LVADs prior to surgery may be enrolled as long as no presurgery immunosuppressives (see list in Appendix B) were administered.]
* Women lactating, pregnant, or of childbearing potential, not using, or who are unwilling to use two reliable forms of contraception simultaneously during the study.
* Men who are not using a reliable contraceptive method
* History of a psychological illness or condition which would interfere with the patient's ability to understand the requirements of the study
* White blood cell count ≤ 2500/mm3, or platelets ≤ 50,000/mm3, or hemoglobin ≤ 6g/dL
* HIV-1, HTLV-1, chronic Hepatitis B, or chronic Hepatitis C infection
* Documented or strong suspicion for pre-operative active infection that has not yet been adequately treated with the recommended course of antimicrobial therapy
* Presence of any chronic myelosuppressive disease or agent that has resulted in either chronic leucopenia or chronic thrombocytopenia
* Active peptic ulcer disease
* Patients who have received within the past 30 days or require concomitant treatment with other investigational drugs (except for those listed in section 8.6 "Concomitant treatment") or immunosuppressive medications that are prohibited for this study (Appendix B)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-11; Primary Completion 2013-11 (Estimated); Study Completion 2018-01-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars-Sinai Medical Center, Beverly Hills, California, United States